CLINICAL TRIAL: NCT02724384
Title: A Multi-Center Pilot Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of the Plasma Treatment System in Improving the Appearance of Onychomycosis
Brief Title: Evaluating the Safety, Tolerability and Preliminary Efficacy of Plasma in Improving the Appearance of Onychomycosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moe Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OM-0030
Record Dates: First submitted 2016-03-22; First posted 2016-03-31 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

ARMS (3):
- Group 1 (Experimental): Plasma treatment using Plasma delivery system A 3 treatments/week for 2 weeks, then monthly
  Interventions: Device: MOE Plasma Delivery System A
- Group 2 (Experimental): Plasma treatment using Plasma delivery system A 2 treatments/week for 2 weeks, then monthly
  Interventions: Device: MOE Plasma Delivery System A
- Group 3 (Experimental): Plasma treatment using Plasma delivery system B 3 treatments/week for 2 weeks, then monthly
  Interventions: Device: MOE Plasma Delivery System B

INTERVENTIONS:
Device: MOE Plasma Delivery System A — Plasma treatment
  Arms: Group 1; Group 2
Device: MOE Plasma Delivery System B — Plasma treatment
  Arms: Group 3

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of using electrical plasma to treat toenail fungus.

DETAILED DESCRIPTION:
75 patients will be recruited at several sites. Patients will be split into 3 groups that have different treatment doses. Patient participation in the study will last 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be between 18 and 70 years of age inclusive, of either sex, and of any race;
2. Subject must have distal subungual infection that affects approximately 25% to 60% of at least one great toenail
3. Dermatophyte infection or infection with C. Albicans in the target great toenail confirmed by identification of a dermatophyte organism in culture;
4. Subject must have at least 3 mm from the proximal end of the target toenail free of infection;
5. Subject must have a target toenail that is assessed as capable of growing approximately 1 mm/month, (e.g., the subject needs to report cutting his or her toenails at least once per month);
6. Subject must be willing to give written informed consent and able to adhere to procedures and visit schedules;
7. Subject must consent to having the toenails photographed during the study period;
8. Woman of childbearing potential: If currently sexually active, must agree to use a medically accepted method of contraception while receiving protocol-specified medication and for 30 days after stopping the study treatments; If not currently active, must agree to use medically accepted method of contraception should she become sexually active during study participation. Methods include condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed intrauterine device, oral or systemic hormonal contraceptive (plus an additional reliable barrier method), and surgical sterilization (e.g., hysterectomy or tubal ligation);
9. Woman of childbearing potential must have a negative serum or urine pregnancy test prior to start of study.

Exclusion Criteria:

1. Subject with more than 6 infected toenails
2. Subject with fingernail onychomycosis
3. Subject with one or more of the following conditions on the primary target toenail:

   1. white superficial onychomycosis
   2. dermatophytoma or "yellow spike/streak"
   3. primarily lateral or bi-lateral disease
   4. toenail thickness greater than 3 mm
   5. inability to become normal in the opinion of the investigator
4. Subject with psoriasis, pincer nail, prior nail surgery, severe moccasin-type tinea pedis requiring treatment, symptomatic interdigital tinea pedis, lichen planus, or other abnormalities that could result in a clinically abnormal nail;
5. Subject with peripheral vascular disease or peripheral circulatory impairment;
6. Subject with uncontrolled diabetes mellitus, subjects with diabetes controlled by insulin or with known diabetic peripheral neuropathy
7. Subject with any known immunodeficiency;
8. Any pacemakers, or any metallic implants or prostheses in the vicinity of the treatment site (such as ankle, foot, etc.);
9. Subject with any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with study evaluations or optimal participation in the study;
10. Subject who has received systemic antifungal therapy within 6 months (except single diflucan tablet for vaginal candida) or topical antifungal therapy applied to the foot or toenails within 1 month of study entry;
11. Subject who has received radiation therapy, chemotherapy, and/or immunosuppressive drugs within 6 months of study, and/or oral corticosteroids for >1 month within the 6 months of study (exception: inhaled steroids);
12. Subject known to have received treatment with investigational drugs or devices within 30 days prior to enrollment into this study;
13. Subject who is unwilling to abstain from any cosmetic nail or foot treatments outside those provided by the study clinic, beyond basic nail trimming (i.e. no spa foot treatments, no pedicures/toenail polish use, no other topical prescription toenail medication);
14. Woman who is breastfeeding, pregnant, or intends to become pregnant (check via urine test only);
15. Subject who is part of the staff personnel directly involved with this study or a family member of the investigational study staff;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with treatment-related adverse events as assessed by CTCAE v4.0 | 12 months
  The primary objective of this study is to compare the short-term safety and tolerability of application of non-ablative electrical plasma to human nails among the different dosing regimes.

SECONDARY OUTCOMES:
Efficacy as assessed by Clinical, Mycological and Complete Cure Rates assessed in accordance with FDA Guidance for onychomycosis trials issued March 7, 2016 | 12 months
  The secondary objective of this study is to evaluate the preliminary efficacy of non-ablative electrical plasma in improving the appearance and treatment of onychomycosis.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - MOE Medical Devices Site 5, Quincy, Massachusetts
  - MOE Medical Devices Site 4, Philadelphia, Pennsylvania
  - MOE Medical Devices Investigational Site 3, Pittsburgh, Pennsylvania
  - MOE Medical Devices Site 6, Austin, Texas
  - MOE Medical Devices Investigational Site 1, College Station, Texas
  - MOE Medical Devices Investigational Site 2, McAllen, Texas
  - MOE Medical Devices Site 7, San Antonio, Texas